CLINICAL TRIAL: NCT03667573
Title: Spinal Excitation to Enhance Mobility in Elderly Adults
Brief Title: Spinal Excitation to Enhance Mobility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E2874-P; I21RX002874 (NIH)
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Aging
Keywords: aging; walking; spinal cord; electrical stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four different parallel groups
Who Masked: Participant
Masking Description: Participants will be masked to the dosage of transcutaneous spinal direct current stimulation (tsDCS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tsDCS Dosage A and textured insoles (Experimental): tsDCS dosage "A" and textured shoe insoles
  Interventions: Device: tsDCS Dosage (A); Other: textured shoe insoles
- tsDCS Dosage B and textured insoles (Experimental): tsDCS dosage "B" and textured shoe insoles
  Interventions: Device: tsDCS Dosage (B); Other: textured shoe insoles
- tsDCS Dosage A and smooth insoles (Experimental): tsDCS dosage "A" and smooth shoe insoles
  Interventions: Device: tsDCS Dosage (A)
- tsDCS Dosage B and smooth insoles (Experimental): tsDCS dosage "B" and smooth shoe insoles
  Interventions: Device: tsDCS Dosage (B)

INTERVENTIONS:
Device: tsDCS Dosage (A) — mild electrical stimulation delivered to lumbosacral spinal cord
  Arms: tsDCS Dosage A and smooth insoles; tsDCS Dosage A and textured insoles
Device: tsDCS Dosage (B) — mild electrical stimulation delivered to lumbosacral spinal cord
  Arms: tsDCS Dosage B and smooth insoles; tsDCS Dosage B and textured insoles
Other: textured shoe insoles — textured shoe insoles
  Arms: tsDCS Dosage A and textured insoles; tsDCS Dosage B and textured insoles

SUMMARY:
Older adults with compromised walking ability have higher rates of morbidity and mortality, more hospitalizations, poorer quality of life, and are less likely to remain independent in the community. It is known that age-related changes in brain and peripheral nerves contribute to loss of walking ability. However, there is a lack of research into how the aging spinal cord affects walking. In older adults, the spinal cord is less excitable, conducts signals more slowly, and is subject to neural noise. Intervening on age-related impairment of the spinal cord to improve walking ability is a very promising but untapped area of research.

DETAILED DESCRIPTION:
It is well known that age-related impairments of the brain and peripheral nerves contribute to a decline in walking function. Age-related impairment of the spinal cord is also a likely contributing factor, as the literature describes a variety of changes in spinal cord structure and function with aging. Specifically, the elderly spinal cord is less excitable, conducts signals more slowly, and is subject to neural noise. Therefore, the investigators are initiating a new line of research with the goal of enhancing walking function in older adults by intervening on age-related neural impairment of the spinal cord. The objective of the proposed study is to establish the feasibility, preliminary efficacy, and variance of response for using transcutaneous spinal direct current stimulation (tsDCS) and textured shoe insoles to excite spinal locomotor circuits and enhance practice-related performance and retention on an obstacle walking task. Enhanced practice and retention effects will support future efforts to translate this approach into a longer term rehabilitation intervention.

Excitatory tsDCS is a non-invasive neuromodulation approach in which a relatively weak electrical current is delivered to the desired region of the spinal cord via electrodes placed on the skin. The electrical current does not cause discharge of action potentials, but rather is designed to bring neurons closer to their discharge threshold by inducing a sub-threshold depolarization of membrane potentials. When combined with a behavioral task, tsDCS has the potential to upregulate neural circuits in a task-specific manner and promote Hebbian neuroplasticity ('fire together, wire together'). The investigators will use a previously established electrode montage to deliver excitatory tsDCS to the lumbosacral spinal cord during practice of a complex obstacle walking task. The investigators also propose to combine the use of textured shoe insoles with tsDCS. This combinatorial approach may be a potent strategy for simultaneously optimizing spinal responsiveness to input from both descending and ascending excitatory signals to spinal centers of locomotor control. The investigators propose a parallel groups study design in which 40 older adults who have walking deficits and who demonstrate a compensatory executive locomotor control strategy will be randomized into one of four groups: 1) dosage "A" tsDCS with smooth insoles (active/smooth); 2) dosage "B" tsDCS with smooth insoles (sham/smooth); 3) dosage "A" tsDCS with textured insoles (active/textured); and 4) dosage "B" tsDCS with textured insole (sham/textured). Participants will be blinded to group assignment. While receiving stimulation, participants will engage in walking practice over a standardized obstacle course. Immediately prior to and following the practice, each participant will be assessed while walking over the course. Practice-related gains in performance will be quantified primarily by fastest safe walking speed. Retention of performance gains will also be assessed at a separate later visit. Intervening on age-related impairment of the spinal cord to improve walking function is a promising but untapped area of research. The proposed intervention techniques are low cost and translatable to real-world settings, which enhances the potential long term impact of this work on the well-being of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Preferred 10m walking speed < 1.0 m/s
* Intact tactile sensation based on two-point discrimination
* Willingness to be randomized to either intervention and to participate in all aspects of study assessment and intervention

Exclusion Criteria:

* Diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition

  * spinal cord injury
  * Alzheimer's
  * Parkinson's
  * stroke, etc.
* Contraindications to non-invasive spinal stimulation including any prior spinal surgical procedure
* Chronic lower back pain
* Obesity, defined as Body Mass Index exceeding 30.

  * This is due to the potential influence of body fat on the amplitude of electrical current flow to the spinal cord.
* Use of medications affecting the central nervous system including, but not limited to:

  * benzodiazepines
  * anti-cholinergic medication and GABAergic medication
* Severe arthritis, such as awaiting joint replacement
* Current cardiovascular, lung or renal disease
* Diabetes
* Terminal illness
* Myocardial infarction or major heart surgery in the previous year
* Cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis

  * early stage breast or prostate cancer
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Difficulty communicating with study personnel

  * including people who cannot speak English
* Uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* Bone fracture or joint replacement in the previous six months
* Current participation in physical therapy for lower extremity function or cardiopulmonary rehabilitation
* Current enrollment in any clinical trial
* Planning to relocate out of the area during the study period
* Clinical judgment of investigative team

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Clark, DSc, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset will be created and shared pursuant to a Data Use Agreement appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The Limited Dataset will be available after the study is completed.

REFERENCES:
- [Result] Clark DJ, Hawkins KA, Winesett SP, Cox BA, Pesquera S, Miles JW, Fuller DD, Fox EJ. Enhancing Locomotor Learning With Transcutaneous Spinal Electrical Stimulation and Somatosensory Augmentation: A Pilot Randomized Controlled Trial in Older Adults. Front Aging Neurosci. 2022 Mar 2;14:837467. doi: 10.3389/fnagi.2022.837467. eCollection 2022. PMID 35309891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study advertisements were mailed to patients of the North Florida/South Georgia Veterans Health System using a mailing list generated by the VA Informatics and Computing Infrastructure. Inclusion criteria for recruitment mailings included age 65 or greater, primary residence in a local zip code, and absence of major medical conditions (based on ICD-9/ICD-10 codes). A screening questionnaire was used to interview individuals by telephone prior to scheduling an onsite screening visit.
Pre-assignment Details: Participants were excluded if they had major health conditions that would affect their safety in the study and/or their ability to perform the study procedures (e.g., ability to walk independently). Other exclusion criteria were excessive body mass index, major somatosensory impairment of the feet, and use of medications affecting the central nervous system.
Period: Overall Study
Arm/Group | tsDCS Dosage A and Textured Insoles | tsDCS Dosage B and Textured Insoles | tsDCS Dosage A and Smooth Insoles | tsDCS Dosage B and Smooth Insoles
Started | 6 | 5 | 5 | 7
Completed | 6 | 5 | 5 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tsDCS Dosage A and Textured Insoles | tsDCS Dosage B and Textured Insoles | tsDCS Dosage A and Smooth Insoles | tsDCS Dosage B and Smooth Insoles | Total
Number analyzed (Participants) | 6 | 5 | 5 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (7.7) | 77.2 (9.9) | 75.8 (5.8) | 79.3 (7.5) | 77.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2 | 4
  Male | 5 | 5 | 4 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 5 | 5 | 7 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Corrected walking speed [Mean (Standard Deviation); unit: meters/second] | 0.850 (.478) | .887 (.272) | .819 (.388) | .913 (.591) | .871 (.435)

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed Change From Baseline
Description: Fastest safe walking speed over the complex walking course (measured as changed between the baseline and follow-up sessions)
Time Frame: Measured at session 2 (2 days after the baseline session)
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | tsDCS Dosage A and Textured Insoles | tsDCS Dosage B and Textured Insoles | tsDCS Dosage A and Smooth Insoles | tsDCS Dosage B and Smooth Insoles
Number analyzed (Participants) | 6 | 5 | 5 | 7
meters/second | .054 (.054) | .078 (.04) | .085 (.04) | .039 (.12)

2. Secondary Outcome: Prefrontal fNIRS Change From Baseline
Description: Prefrontal brain activity while walking at fastest safe walking speed over the complex walking course (measured by fNIRS as change between baseline and follow-up session)
Time Frame: Measured at session 2 (2 days after the baseline session)
Measure: Mean (Standard Deviation); unit: microMolar
Arm/Group | tsDCS Dosage A and Textured Insoles | tsDCS Dosage B and Textured Insoles | tsDCS Dosage A and Smooth Insoles | tsDCS Dosage B and Smooth Insoles
Number analyzed (Participants) | 6 | 5 | 5 | 7
microMolar | -1.21 (0.93) | 0.24 (1.15) | 0.14 (0.47) | 0.17 (0.62)

ADVERSE EVENTS:
Time Frame: 3 days
Description: An adverse event is any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's involvement in the research, whether or not considered related to participation in the research.
Arm/Group | tsDCS Dosage A and Textured Insoles | tsDCS Dosage B and Textured Insoles | tsDCS Dosage A and Smooth Insoles | tsDCS Dosage B and Smooth Insoles
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03667573/Prot_SAP_000.pdf